CLINICAL TRIAL: NCT06975709
Title: ASSOCIATION BETWEEN TEMPOROMANDIBULAR DISORDERS AND SLEEP DISORDERS
Acronym: Gnathology TMD
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Luigi Ferini Strambi, Prof, IRCCS San Raffaele
Other Study IDs: IRCCS San Raffaele Hospital; CET 49-2025 (Registry Identifier: CET Lombardia 1)
Record Dates: First submitted 2025-03-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Temporomandibular Disorders (TMD); Sleep
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with TMD: Temporomandibular disorder (TMD), a common cause of chronic orofacial pain, is a group of painful and/or dysfunctional conditions of the masticatory muscles, temporomandibular joint (TMJ) and associated structures.
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — The diagnostic questionnaires will be administered and the participants' responses will subsequently be analyzed, evaluating the presence of temporomandibular disorders (DTMs) in patients with sleep disorders.
  The questionnaires will be administered to patients with a previous diagnosis of sleep disorder carried out at a specialist centre, consecutively belonging to the outpatient clinics of both centers U.O of Neurology-Sleep Disorders Center and U.O of Dentistry.

SUMMARY:
ASSOCIATION BETWEEN TEMPOROMANDIBULAR DISORDERS AND SLEEP DISORDERS

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are complex conditions, which can have a significant impact on patients' health and quality of life. Furthermore, they are unclearly associated with sleep disorders. The aim of the study is to investigate the prevalence of TMD in patients with sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Famale and Male
* Signature of the privacy information form
* Signature of the informed consent form of the protocol
* Subjects capable of understanding and wanting
* Subjects suffering from a sleep disorder (Insomnia,Hypersomnia,Restless legs syndrome,REM sleep behavior disorder,Narcolepsy,Obstructive sleep apnea syndrome (OSAS),Primary snoring, REM parasomnias,Nocturnal epilepsy)

Exclusion Criteria:

* Physical trauma to the head and neck area
* Painful oral pathologies (e.g. pulpitis, tooth fractures, tooth abscesses, tooth decay, canker sores and mucosal wounds)
* Recent dental treatments that may cause pain (e.g. tooth extraction, tooth root canal)
* Use of oral contraceptives
* Subjects not capable of understanding and wanting
* Patients suffering from neurological pathologies that may interfere with the completion of the questionnaires (ES dementia) or psychiatric pathologies or drug use as per DSM-5 criteria (including schizophrenia, bipolar, major depression, substance abuse, personality disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population must include Female and Male over 18 y.o with sleep disorders that meet inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | at enrollment
  The main aim of the present study is to evaluate the prevalence of TMDs in patients with sleep disorders. This population was selected in order to contribute, in the context of scientific research, to the investigation into the association between temporomandibular disorders and sleep disorders, which include all those disorders that compromise both the quantity and quality of sleep with repercussions important on general health and quality of life, like:
  * Insomnia
  * Hypersomnia
  * Restless legs syndrome
  * REM sleep behavior disorder
  * Narcolepsy
  * Obstructive sleep apnea syndrome (OSAS)
  * Primary snoring
  * REM parasomnias (Sleepwalking, arousal disorders, excessive daytime sleepiness and night terrors)
  * Nocturnal epilepsy Patients with sleep disorders may be recruited in the observational study conducted by the University's Department of Dentistry Vita-Salute San Raffaele and the Neurology-sleep disorders unit of the San Raffaele Hospital in Turro, aimed at evaluating the prevalence of T

SECONDARY OUTCOMES:
Secondary Outcome | at enrollment
  Through this study we also want to evaluate the difference between the prevalence of TMDs in patients with sleep disorders and the prevalence of TMDs in non-patological population through the data present in the scientific literature.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS San Raffaele Hospital, Milan, Italy
  - IRCCS Ospedale San Raffaele Turro, Milan, Milano